CLINICAL TRIAL: NCT04596345
Title: Psychological Distress in Emerging Adulthood: A Longitudinal Study
Acronym: DistressEA
Status: Completed | Type: Observational
Sponsor: Universidad de las Americas - Quito (Other)
Responsible Party: Principal Investigator, Clara Paz, Researcher, Universidad de las Americas - Quito
Other Study IDs: PSI.CPE.20.01
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Psychological Distress
Keywords: Young Adult; Life Change Events; Students; Mental Health; Observational Study; Longitudinal Studies; Surveys and Questionnaires; Self Report
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- University students: This group will include all those participants who declare to be attending a study program to get a higher education degree.
  No intervention will be applied.
- Non-university-attending peers: This group will include all those participants who are not attending a study program to get a higher education degree.
  No intervention will be applied.

SUMMARY:
Emerging adulthood (18-29 years) is a critical stage in lifespan development. During this stage, people experience instability: shifts from their families of origin, breakups of relationships and job changes are frequent before most young adults stabilize their lives and make more lasting decisions. This study seeks to understand the psychological distress of emerging adults in Quito, Ecuador and define how it varies over a year.

DETAILED DESCRIPTION:
Emerging adulthood is often a period of some instability with relationship changes and often a series of job changes before life trajectories clarify and more lasting decisions are possible. These changes often produce distress and they might explain why most of the symptoms that impact the individual's mental health throughout their lives appear at this stage, although full-blown disorders are often only diagnosed subsequently. There are several studies that describe the prevalence of mental disorders in this age group, however, there are few studies that refer to how psychological distress changes during this phase of emotional, social, and financial instability. The few existent studies refer mostly to college student populations, with relative neglect of the non-student populations.

The objective of this study is to analyze the intraindividual changes in psychological distress of emerging adults over one year. These changes will be compared between those participants who are college students and those who are not. Sociodemographic data will be recorded in the first assessment and the last assessment, while psychological distress and health-related quality of life will be monitored bimonthly for seven assessment points in total. Everyday relevant events will be also recorded bimonthly for seven assessment points, and this information will be used as a time-varying covariate. An electronic survey will be used for data collection through formr system (https://formr.org/).

The results of this research will show if the distress changes significantly in the studied population for one year and it will be possible to identify some of the events and variables that are related to these changes. This knowledge might help to create interventions that are tailored to the needs of this population.

ELIGIBILITY:
Inclusion Criteria:

* Competence to read and understand Spanish
* Living in Ecuador
* Being a student (for the student cohort)
* Not attending to a formal student program (for the non-student cohort)

Exclusion Criteria:

* None

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population will be emerging adults from Ecuador students and non-students as one objective is to compare psychological distress variability between both populations.
Sampling Method: Non-Probability Sample
Enrollment: 1168 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change on the Clinical Outcomes in Routine Evaluation (CORE) | One year (seven assessment points at two-month intervals)
  A 34-item self-reported measure that assess psychological distress and how it changes considering four dimensions: subjective well-being (four items), problems and or symptoms (twelve items), life function (twelve items) and risk to self and others (six items). Higher scores indicate higher psychological distress. It is measure that can be downloaded free of charge from: www.coresystemtrust.org.uk. The Clinical Outcomes in Routine Evaluation- Outcome Measure(CORE-OM) has shown good psychometric properties in college students (and a non-student general population sample) from Ecuador (http://dx.doi.org/10.1186/s40359-020-00443-z)

SECONDARY OUTCOMES:
EuroQol five-dimensions - three-level (EQ-5D-3L) | One year (seven assessment points at two-month intervals)
  A 5-item self-report measure of health-related quality of life states in adults, considering five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & Depression), each of which has three severity levels that are described by statements appropriate to that dimension. As result a 5-digit number describes person's health state profile. Higher scores represent more problems with regard to each dimension.
EuroQol Visual Analogue Scale (EQ VAS) | One year (seven assessment points at two-month intervals)
  This scale records the patient's self-rated health on a vertical visual analogue scale that ranges from 0= 'Best imaginable health state' to 100 = 'Worst imaginable health state'. The VAS will be used as a quantitative measure of health outcome .

CONTACTS AND LOCATIONS:
Locations (1):
- Metropolitan District, Quito, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paz C, Evans C. A comparison of mental health of student and not student emerging adults living in Ecuador. Sci Rep. 2023 Jan 27;13(1):1487. doi: 10.1038/s41598-023-27695-0. PMID 36707675
- [Derived] Paz C, Osejo-Taco G, Evans C. Trajectories of success and/or distress: protocol for an observational cohort study investigating changing psychological distress among emerging Ecuadorian adults over a year. BMJ Open. 2021 Dec 20;11(12):e056361. doi: 10.1136/bmjopen-2021-056361. PMID 34930747

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT04596345/SAP_001.pdf